CLINICAL TRIAL: NCT04591015
Title: Dulce Digital-COVID Aware (DD-CA) Discharge Texting Platform for US/Mexico Border Hispanics With Diabetes + COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Athena Philis-Tsimikas, Corporate Vice President, Scripps Whittier Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3R01DK112322-05S1 (NIH); 3R01DK112322-05S1 (NIH)
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2; Covid19
Keywords: Type 2 Diabetes; COVID-19
MeSH Terms: conditions — Diabetes Mellitus, Type 2; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DD-CA (Experimental): In the DD-CA arm, participants will be offered a proven digital texting platform in their language of preference (Spanish/English) as part of the diabetes transitions discharge program with added COVID support messages.
  Interventions: Behavioral: Hospital: DD-CA
- Usual Care (UC) (Active Comparator): UC participants will not receive the added COVID support messages, both arms will have a referral placed to the Diabetes Transitions Service (DTS) as part of usual care at the time of discharge.
  Interventions: Behavioral: Hospital: Usual Care (UC)

INTERVENTIONS:
Behavioral: Hospital: DD-CA — In the DD-CA group, participants will be offered a proven digital texting platform in their language of preference (Spanish/English) as part of the diabetes transitions discharge program with educational, motivational and medication adherence messaging that is currently an arm of our parent DD-ME grant with added COVID support messages that provide information addressing identified barriers in Hispanic underserved communities (e.g. obtaining testing supplies and medications, accessing routine medical care, and completing other important diabetes self-management behaviors such as healthful eating, exercise, social distancing, quarantine, and stay-at-home/lockdown guidelines).
  Arms: DD-CA
Behavioral: Hospital: Usual Care (UC) — In the UC group, participants will not receive the added COVID support messages, both groups will have a referral placed to the Diabetes Transitions Service (DTS) at the time of discharge as part of usual care. Participants will be contacted by a peer health coach following protocol to coordinate care with outpatient health and other community resources.
  Arms: Usual Care (UC)

SUMMARY:
The COVID-19 pandemic has triggered extremely high hospitalization rates where mitigation strategies are urgently necessary to aid vulnerable Hispanic and Latino populations who are experiencing health disparities as well as high type 2 diabetes (T2D) prevalence with poor clinical outcomes when compared to non-Hispanic populations. The supplemental Dulce Digital-COVID Aware (DD-CA) intervention addresses specific barriers in diverse underserved Hispanic and Latino communities to improve glucose control and lower transmission of COVID-19 during a highly vulnerable period post hospitalization discharge, to reduce hospital readmission rates. This supplement will integrate COVID educational messaging with glucose management messaging within a low-cost, easily adoptable digital texting platform and offer critical information in a culturally and linguistically relevant manner to address specific barriers in diverse underserved communities.

DETAILED DESCRIPTION:
Hispanics, a group that shows higher type 2 diabetes (T2D) prevalence, and poor self-management and clinical outcomes, have been disproportionally adversely impacted by COVID-19. The California Department of Public Health reports that Hispanics make up 39% of California's population but an unprecedented 57% of the confirmed COVID-19 cases. This devastating finding is especially notable on the US/Mexico border. Diabetes has emerged as a leading risk factor for severe COVID-19 illness leading to hospitalization, is associated with greater disease severity and mortality and is an independent predictor of intensive care placement and invasive ventilation. It is becoming increasingly clear that maintaining good glucose control improves prognosis of COVID-19 among people with pre-existing T2D. However, social distancing, quarantine, and stay-at-home/lockdown guidelines may impact one's ability to maintain adequate glycemic control. Research is needed to evaluate the effect and clinical outcomes of a flexible, easily adopted low cost digital intervention that improves glucose excursions and provides urgently needed COVID-19 mitigation strategies, among rapidly rising groups of high-risk Hispanics with poorly controlled T2D in US/Mexico border communities. Strong evidence from our parent grant Dulce Digital-Me (DD-ME), supports the use of technology (such as text messaging) alone or in combination with coaching interventions as a viable and desired method of delivering tailored diabetes self-management education and COVID awareness messaging to high-risk, underserved populations in a manner that is more convenient for both patients and staff while having the added benefit of being cost-effective for health systems, especially within low resource settings. However, effective interventions may encounter barriers which preclude guaranteed success upon implementation in the real world. This project, taking place along the San Diego/Tijuana border, historically the busiest land port of entry in the Western Hemisphere, will assess the effect of providing an enhanced digital texting intervention-Dulce Digital-COVID Aware (DD-CA) to N = 172 Hispanic patients with T2D upon discharge from a recent hospitalization. Key outcomes will assess the impact of DD-CA on hospital readmissions at 30, 90 and 180 days post-discharge, glucose control and patient reported outcomes at 90 and 180 days post-discharge while also assessing COVID status and the implementation process. Given that DD-CA offers the potential to address many of the practical barriers to access and extend the reach of diabetes services, while additionally providing COVID awareness support, it offers an ideal low-cost and flexible solution to reduce hospital admissions and re-admissions in US/Mexico border communities significantly and simultaneously affected by COVID-19 and T2D. Implemented in a typical hospital and post-discharge setting, it augments existing care team processes, thus providing a valuable test of real-world effectiveness. More importantly, by helping to reduce existing inequities in access to diabetes and COVID-19 care, this program aims to improve health outcomes on a larger scale.

ELIGIBILITY:
Inclusion Criteria:

* Are a patient admitted to a Scripps Mercy Hospital,
* Consider yourself Hispanic/Latino, of any race
* Are 18 years of age or older,
* Speak English or Spanish,
* Have type 2 diabetes and A1c ≥ 7% in the last 90 days, and
* Have a cellphone that can receive/send text messages.

Exclusion Criteria:

* Are pregnant,
* Are currently participating in another diabetes or COVID-19 related study, or
* Do not meet all eligibility inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athena Philis-Tsimikas, MD, Principal Investigator — Scripps Whittier Diabetes Institute
Locations (1):
- Scripps Mercy Hospital Chula Vista, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DD-CA | Usual Care (UC)
Started | 86 | 86
Completed | 58 | 68
Not Completed | 28 | 18
Not completed — Death | 6 | 4
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 16 | 11

BASELINE CHARACTERISTICS:
Population: Patients of a hospital in South San Diego County that serves mostly Hispanic/Latino, low income and poorly managed type 2 diabetes.
Groups:
- Total: Total of all reporting groups
Arm/Group | DD-CA | Usual Care (UC) | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.23 (14.20) | 61.33 (11.24) | 57.78 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 48 | 83
  Male | 51 | 38 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 86 | 86 | 172
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 8
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 37 | 32 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 46 | 49 | 95
Region of Enrollment [Number; unit: participants]
  United States | 86 | 86 | 172
Les than High School Education [Count of Participants; unit: Participants] | 41 | 39 | 80
Income Less than 30,000 per year [Count of Participants; unit: Participants] | 58 | 60 | 118
Not Employed [Count of Participants; unit: Participants] | 58 | 66 | 124
Married or Cohabitating [Count of Participants; unit: Participants] | 49 | 46 | 95
Born in Mexico [Count of Participants; unit: Participants] | 61 | 58 | 119
Primary Language is Spanish [Count of Participants; unit: Participants] | 63 | 59 | 122
Has Some Type of Health Insurance [Count of Participants; unit: Participants] | 66 | 78 | 144
Cardiometabolic Conditions [Count of Participants; unit: Participants] | 86 | 86 | 172
Hospital Visit Length of Stay in Days [Mean (Standard Deviation); unit: days] | 7.02 (6.64) | 5.45 (3.92) | 6.24 (5.50)
Diabetes Distress Scale [Mean (Standard Deviation); unit: units on a scale] | 1.85 (0.85) | 1.93 (0.86) | 1.89 (0.86)
Summary of Diabetes Self-Care Activities - Diet [Mean (Standard Deviation); unit: units on a scale] | 4.15 (1.92) | 4.20 (1.62) | 4.18 (1.78)
Summary of Diabetes Self-Care Activities - Excercise [Mean (Standard Deviation); unit: units on a scale] | 2.72 (2.90) | 2.38 (2.96) | 2.55 (2.92)
Summary of Diabetes Self-Care Activities - Blood glucose testing [Mean (Standard Deviation); unit: units on a scale] | 2.88 (3.21) | 4.13 (3.12) | 3.51 (3.21)
Patient Reported Outcomes Measurement Information System Global-10 Health Scale - Physical Health [Mean (Standard Deviation); unit: units on a scale] | 12.41 (3.25) | 11.98 (3.23) | 12.19 (3.24)
Patient Reported Outcomes Measurement Information System Global-10 Health Scale - Mental Health [Mean (Standard Deviation); unit: units on a scale] | 13.50 (3.09) | 13.31 (3.27) | 13.40 (3.18)

OUTCOME MEASURES:

1. Primary Outcome: Hospital Readmission Rate Within 30 Days of Discharge
Description: Number of Participants With at Least 1 Hospital Readmission Within 30 Days After Enrollment, analyzed for full study sample
Time Frame: Within 30 days of discharge
Measure: Count of Participants; unit: Participants
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 86 | 86
Participants | 24 | 13
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.0626, Fisher Exact

2. Primary Outcome: Glycosylated Hemoglobin (HbA1c) - Change From Baseline to 90 Days
Description: Change in Glycosylated Hemoglobin (HbA1c) 90 days from baseline. A negative mean indicates positive change in HbA1c.
Time Frame: 90 days from baseline
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 27 | 29
percentage of HbA1c | -2.69 (2.53) | -1.45 (2.04)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Only includes participants who completed a 90-day lab; Test type: Superiority; p = 0.0496, t-test, 2 sided

3. Primary Outcome: Glycosylated Hemoglobin (HbA1c) - Change From Baseline to 180 Days
Description: Change in Glycosylated Hemoglobin (HbA1c) 180 days from baseline. A negative mean indicates positive change in HbA1c.
Time Frame: 180 days from baseline
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 30 | 34
percentage of HbA1c | -2.03 (2.66) | -0.91 (2.02)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Only includes participants who completed a 180-day lab; Test type: Superiority; p = 0.0651, t-test, 2 sided

4. Secondary Outcome: Hospital Readmission Rate Within 90 Days of Discharge
Description: Number of Participants With at Least 1 Hospital Readmission Within 90 Days After Enrollment, analyzed for full study sample.
Time Frame: Within 90 days of discharge
Measure: Count of Participants; unit: Participants
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 86 | 86
Participants | 32 | 30
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.8739, Fisher Exact

5. Secondary Outcome: Diabetes Distress Scale - Change From Baseline to 90 Days
Description: Diabetes distress as reported by patient; 90 days from baseline. The minimum score is 1 and maximum score is 6 with a higher score representing worse outcome or greater diabetes related emotional stress. A negative mean indicates a positive change in the diabetes distress score.
Time Frame: 90 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 53 | 56
score on a scale | -0.42 (0.77) | -0.31 (0.69)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.4702, t-test, 2 sided

6. Secondary Outcome: Diabetes Distress Scale - Change From Baseline to 180 Days
Description: Diabetes distress as reported by patient; 180 days from baseline. The minimum score is 1 and maximum score is 6 with a higher score representing worse outcome or greater diabetes-related emotional stress. A negative mean indicates a positive change in the diabetes distress score.
Time Frame: 180 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 47 | 47
score on a scale | -0.56 (0.68) | -0.35 (0.58)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.1258, t-test, 2 sided

7. Secondary Outcome: Summary of Diabetes Self-Care Activities - Diet - Change From Baseline to 90 Days
Description: Diabetes self-care activities related to Diet as reported by patient; 90 days from baseline; The minimum score is 0 and maximum score is 7 with a higher score representing better adherence to diabetes diet self-management behaviors. A positive mean indicates a positive change in the diet self-care activities.
Time Frame: 90 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 53 | 56
score on a scale | 0.99 (1.99) | 1.06 (1.89)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.8635, t-test, 2 sided

8. Secondary Outcome: Summary of Diabetes Self-Care Activities - Exercise - Change From Baseline to 90 Days
Description: Diabetes self-care activities related to Exercise as reported by patient; 90 days from baseline; The minimum score is 0 and maximum score is 7 with a higher score representing better adherence to diabetes exercise self-management behaviors. A positive mean indicates a positive change in exercise self-care activities.
Time Frame: 90 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 53 | 56
score on a scale | 1.77 (3.41) | 0.47 (3.45)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.0471, t-test, 2 sided

9. Secondary Outcome: Summary of Diabetes Self-Care Activities - Blood Sugar - Change From Baseline to 90 Days
Description: Diabetes self-care activities related to Blood Sugar as reported by patient; 90 days from baseline; The minimum score is 0 and maximum score is 7 with a higher score representing better adherence to diabetes blood sugar self-management behaviors. A positive mean indicates a positive change in blood sugar self-care activities.
Time Frame: 90 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 53 | 56
score on a scale | 3.08 (3.37) | 1.64 (3.11)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.0218, t-test, 2 sided

10. Secondary Outcome: Summary of Diabetes Self-Care Activities - Diet - Change From Baseline to 180 Days
Description: Diabetes self-care activities related to Diet as reported by patient; 180 days from baseline; The minimum score is 0 and maximum score is 7 with a higher score representing better adherence to diabetes diet self-management behaviors. A positive mean indicates a positive change in diet self-care activities.
Time Frame: 180 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 47 | 49
score on a scale | 1.08 (2.08) | 0.82 (1.69)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.5090, t-test, 2 sided

11. Secondary Outcome: Summary of Diabetes Self-Care Activities - Exercise - Change From Baseline to 180 Days
Description: Diabetes self-care activities related to Exercise as reported by patient; 180 days from baseline; The minimum score is 0 and maximum score is 7 with a higher score representing better adherence to diabetes exercise self-management behaviors. A positive mean indicates a positive change in exercise self-care activities.
Time Frame: 180 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 47 | 49
score on a scale | 1.89 (3.41) | 1.33 (3.13)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.4034, t-test, 2 sided

12. Secondary Outcome: Summary of Diabetes Self-Care Activities - Blood Sugar - Change From Baseline to 180 Days
Description: Diabetes self-care activities related to Blood Sugar as reported by patient; 180 days from baseline; The minimum score is 0 and maximum score is 7 with a higher score representing better adherence to diabetes blood sugar self-management behaviors. A positive mean indicates a positive change in blood sugar self-care activities.
Time Frame: 180 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 47 | 49
score on a scale | 2.38 (3.19) | 0.76 (3.41)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.0175, t-test, 2 sided

13. Secondary Outcome: COVID-19 Patient Survey (Phenix Toolkit) Within 90 Days of Discharge
Description: COVID-19 Patient Survey was used to assess COVID-19 diagnosis status and determine whether new infections occurred in the 90-day post-discharge time frame.
Time Frame: Within 90 days of discharge
Measure: Count of Participants; unit: Participants
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 65 | 59
Participants | 5 | 2
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.4435, Fisher Exact

14. Secondary Outcome: COVID-19 Patient Survey (Phenix Toolkit) Within 180 Days of Discharge
Description: COVID-19 Patient Survey was used to assess COVID-19 diagnosis status and determine whether new infections occurred in the 180-day post-discharge time frame.
Time Frame: Within 180 days of discharge
Measure: Count of Participants; unit: Participants
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 54 | 53
Participants | 8 | 4
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.7417, Fisher Exact

15. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 Health Scale - Physical - Change Between Baseline and 90 Days
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 Health Scale was a measure of overall score patient-reported physical health collected at baseline and 90 days. The minimum score on this scale is 0 and maximum score is 100. A higher score indicates a better outcome/higher quality of life. When the means are calculated between baseline and 90 days, a positive mean indicates a better outcome/higher quality of life.
Time Frame: 90 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 54 | 55
score on a scale | 0.87 (2.73) | 0.55 (3.21)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.5779, t-test, 2 sided

16. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 Health Scale - Mental - Change Between Baseline and 90 Days
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 Health Scale was a measure of overall score patient-reported mental health 90 days from baseline. The minimum score on this scale is 0 and maximum score is 100. A higher score indicates a better outcome/higher quality of life. When the means are calculated between baseline and 90 days, a positive mean indicates a better outcome/higher quality of life and a negative mean indicates a worse outcome/lower quality of life.
Time Frame: 90 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 54 | 55
score on a scale | 0.91 (2.74) | -0.16 (2.92)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.0493, t-test, 2 sided

17. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 Health Scale - Physical - Change Between Baseline and 180 Days
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 Health Scale was a measure of overall score patient-reported physical health 180 days from baseline. The minimum score on this scale is 0 and maximum score is 100. A higher score indicates a better outcome/higher quality of life. When the means are calculated between baseline and 180 days, a positive mean indicates a better outcome/higher quality of life.
Time Frame: 180 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 48 | 47
score on a scale | 1.59 (3.33) | 0.38 (3.37)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.0773, t-test, 2 sided

18. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 Health Scale - Mental - Change Between Baseline and 180 Days
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 Health Scale was a measure of overall score patient-reported mental health 180 days from baseline. The minimum score on this scale is 0 and maximum score is 100. A higher score indicates a better outcome/higher quality of life. When the means are calculated between baseline and 180 days, a positive mean indicates a better outcome/higher quality of life, and a negative mean indicates a worse outcome/lower quality of life.
Time Frame: 180 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 48 | 47
score on a scale | 0.81 (3.00) | -0.21 (2.82)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.0921, t-test, 2 sided

19. Secondary Outcome: Knowledge, Attitudes and Practice Toward COVID-19 Survey - Change From Baseline to 90 Days
Description: Knowledge, Attitudes and Practice Toward COVID-19 Survey was used to measure knowledge and attitudes related to COVID-19 at 90 days from baseline. The minimum score on this scale is 0 and maximum score is 12, with higher scores indicating greater knowledge of COVID-19. A negative mean indicates lesser knowledge of COVID-19.
Time Frame: 90 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 55 | 55
score on a scale | -0.64 (1.77) | -0.29 (1.26)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.2404, t-test, 2 sided

20. Secondary Outcome: Knowledge, Attitudes and Practice Toward COVID-19 Survey - Change From Baseline to 180 Days
Description: Knowledge, Attitudes and Practice Toward COVID-19 Survey was used to measure knowledge and attitudes related to COVID-19 at 180 days from baseline. The minimum score on this scale is 0 and maximum score is 12, with higher scores indicating greater knowledge of COVID-19. A negative mean indicates lesser knowledge of COVID-19.
Time Frame: 180 days from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DD-CA | Usual Care (UC)
Number analyzed (Participants) | 48 | 48
score on a scale | -0.48 (1.65) | -0.52 (1.44)
Statistical Analysis 1: Comparison: DD-CA vs Usual Care (UC); Test type: Superiority; p = 0.8955, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 18 months
Description: All cause mortality
Arm/Group | DD-CA | Usual Care (UC)
All-Cause Mortality (participants affected / at risk) | 6/86 | 4/86
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86
Other Adverse Events (participants affected / at risk) | 0/86 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT04591015/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT04591015/ICF_000.pdf